CLINICAL TRIAL: NCT00621530
Title: Effect of Intrathecal Ketorolac on Mechanical Hypersensitivity After Total Hip Arthroplasty
Brief Title: Effect of Spinal Ketorolac on Mechanical Hypersensitivity After a Total Hip Replacement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to discontinuation of Acular PF (investigational medication)
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00004736; 5R37GM048085 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Hip Arthroplasty
Keywords: Total hip arthroplasty; Total hip replacement; Pain, postoperative; Ketorolac; Patients undergoing unilateral total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketorolac (Experimental): ketorolac 2 mg ketorolac tromethamine opthalmic solution
  Interventions: Drug: ketorolac tromethamine opthalmic solution
- Placebo (Placebo Comparator): placebo will be added to the patient's routine spinal anesthetic for surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ketorolac tromethamine opthalmic solution — ketorolac 2 mg will be added to the patient's routine spinal anesthetic for surgery
  Other Names: Acular- Preservative Free (PF); Ketorolac
  Arms: Ketorolac
Drug: placebo — placebo will be added to the patient's routine spinal anesthetic for surgery
  Arms: Placebo

SUMMARY:
Chronic pain in patients following total hip replacement seems to be a significant problem. Previous research has shown that more effective pain management in the early postoperative period may decrease the incidence of the development of chronic pain states.

This study will evaluate whether ketorolac (a non steroidal anti-inflammatory drug) given into the spinal fluid before surgery will reduce the area of sensitivity (or pain to light touch) following surgery. Patients will be monitored during their postoperative hospital stay and then contacted by telephone at 8 weeks and 6 months after surgery and questioned about any pain they are having at their surgical site. Patients that are still experiencing pain at 6 months will be asked to return to the medical center for the study staff to assess their pain or sensitivity at the surgical site.

DETAILED DESCRIPTION:
Surgery results in hypersensitivity to mechanical stimuli surrounding the wound and in a subset of patients, also results in chronic pain. The purpose of the study is to test whether intrathecal ketorolac, by selectively and effectively blocking cyclooxygenase in the spinal cord, will reduce hypersensitivity surrounding the surgical wound in patients with high risk for developing chronic pain after surgery. We have chosen to study patients having total hip arthroplasty (THA) because chronic pain seems to be a significant problem after surgery. We will sample cerebrospinal fluid (CSF) prior to injection of the study medication for subsequent prostaglandin E2 (PGE2) analysis in each patient. We will also assess each patient at 48 hours after their surgery for hypersensitivity at their surgical site.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II, III
* > Age 18
* Primary unilateral total hip arthroplasty under spinal anesthesia

Exclusion Criteria:

* Known allergy to study medication
* Weight > 300 pounds
* Obstructive sleep apnea
* Patients with severe renal (kidney) or hepatic (liver) disease, allergy to ketorolac, amino amide local anesthetic, or contraindications to spinal anesthesia
* Patients on dialysis for kidney failure or patients that are jaundice or have a diagnosis of liver failure
* Patients routinely taking narcotic pain medications for pain other than their primary hip pain
* Patients that are taking Lyrica (pregabalin) or Gabapentin (neurontin) for the treatment of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang L, Bauer M, Curry R, Larsson A, Sessler DI, Eisenach JC. Intrathecal ketorolac does not improve acute or chronic pain after hip arthroplasty: a randomized controlled trial. J Anesth. 2014 Oct;28(5):790-3. doi: 10.1007/s00540-014-1798-6. Epub 2014 Feb 18. PMID 24535482

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac: ketorolac 2 mg
  ketorolac tromethamine opthalmic solution: ketorolac 2 mg will be added to the patient's routine spinal anesthetic for surgery
Period: Overall Study
Arm/Group | Ketorolac | Placebo
Started | 30 | 32
Completed | 28 | 29
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 17 | 31
Region of Enrollment [Number; unit: participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Area of Hypersensitivity to Mechanical Stimuli Surrounding the Wound 48 Hours After Surgery
Description: Hyperalgesia (using a von Frey filament) and allodynia (using a cotton swab) were evaluated around the surgical site 48 hours after surgery.
Time Frame: 48 hours
Population: These are data from the 57 subjects who remained in the study at the time of the primary outcome measure 48 hr after surgery
Measure: Median (Full Range); unit: area in centimeters squared
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 29
area in centimeters squared | 0 [0 to 84] | 0 [0 to 49]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Power calculation assumed that all subjects would have an area of hypersensitivity surrounding the wound at 48 hours. We found that only 1 subject in the placebo group and 3 subjects in the ketorolac group had non-zero areas of hypersensitivity; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0

2. Secondary Outcome: Present Pain Intensity
Description: Pain was assessed preoperatively, 2 days, and 2 and 6 months after surgery using a 0-10 (10 being worse) verbal Present Pain Intensity (PPI) scale
Time Frame: 6 months
Population: Some subjects were missed to follow up at different times
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketorolac: ketorolac tromethamine opthalmic solution, 2 mg added to the patient's routine spinal anesthetic for surgery
- Placebo: sterile saline placebo added to the patient's routine spinal anesthetic for surgery
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 29
units on a scale
  Preoperative | 1.7 (1.5) | 1.6 (1.1)
  Postoperative: 2 days | 2.1 (1.8) | 2.5 (2.3)
  Postoperative: 2 months: number analyzed (Participants) | 28 | 27
  Postoperative: 2 months | 0.6 (1.2) | 0.2 (0.3)
  Postoperative: 6 months: number analyzed (Participants) | 23 | 28
  Postoperative: 6 months | 0.4 (0.6) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.78, ANOVA; Repeated measures ANOVA

3. Secondary Outcome: McGill Pain Intensity
Description: Pain was assessed 2 days and 2 and 6 months after surgery using a validated questionnaire wherein subjects rate the degree to which adjectives describe the intensity of their pain experience. This is termed the McGill Pain Intensity Score and is scored from 0 to 33 with 33 being the highest pain intensity.
Time Frame: 6 months
Population: Some subjects were missed to follow up at different times
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 29
units on a scale
  Postoperative: 2 days | 11 (6.3) | 10 (6.6)
  Postoperative: 2 months: number analyzed (Participants) | 28 | 27
  Postoperative: 2 months | 2.3 (3.3) | 3.1 (4.1)
  Postoperative: 6 months: number analyzed (Participants) | 23 | 28
  Postoperative: 6 months | 1.4 (3.8) | 1.2 (2.2)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.87, ANOVA; Repeated measures ANOVA

4. Secondary Outcome: McGill Affective Pain
Description: Pain was assessed 2 days, and 2 and 6 months after surgery using a validated questionnaire wherein subjects rate the degree to which adjectives describe the emotional component of their pain experience. This is termed the McGill Pain Affective Score and is scored from 0 to 12 with 12 being the highest pain emotional impact.
Time Frame: 6 months
Population: Some subjects were missed to follow up at different times
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 29
units on a scale
  Postoperative: 2 days | 2.3 (2.5) | 2.3 (2.5)
  Postoperative: 2 months: number analyzed (Participants) | 28 | 27
  Postoperative: 2 months | 0.4 (0.8) | 0.5 (0.8)
  Postoperative: 6 months: number analyzed (Participants) | 23 | 28
  Postoperative: 6 months | 0.1 (0.8) | 0.4 (0.8)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.66, ANOVA; Repeated measures ANOVA

5. Secondary Outcome: Neuropathic Pain Symptom Inventory
Description: Pain was assessed 2 days, and 2 and 6 months after surgery using a validated questionnaire to assess the degree of neuropathic characteristics of pain. This is termed the Neuropathic Pain Symptom Inventory which is scored 0-100 with 100 being the worst possible pain.
Time Frame: 6 months
Population: Some subjects were missed to follow up at different times
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketorolac: ketorolac tromethamine opthalmic solution 2 mg added to the patient's routine spinal anesthetic for surgery
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 29
units on a scale
  Postoperative: 2 days | 13 (13) | 21 (14)
  Postoperative: 2 months: number analyzed (Participants) | 28 | 27
  Postoperative: 2 months | 2.9 (4.6) | 4.5 (7.2)
  Postoperative: 6 months: number analyzed (Participants) | 23 | 28
  Postoperative: 6 months | 2.4 (6.6) | 1.4 (3.2)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.83, ANOVA; Repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ketorolac | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

LIMITATIONS AND CAVEATS:
The trial was terminated because the study drug became unavailable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-02-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT00621530/Prot_SAP_000.pdf
  • Informed Consent Form (2009-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT00621530/ICF_001.pdf